CLINICAL TRIAL: NCT05353673
Title: The Combination of Sitagliptin and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia: A Randomized, Controlled, Multicenter, Open-label Trial
Brief Title: The Combination of Sitagliptin and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-ITP035
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Immune Thrombocytopenia; Blood Coagulation Disorders; Thrombocytopenia; Physiological Effects of Drugs
Keywords: Sitagliptin; Immune Thrombocytopenia; Danazol
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Coagulation Disorders; Thrombocytopenia | interventions — Sitagliptin Phosphate; Danazol

STUDY DESIGN:
Intervention Model Description: The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 100 adults with steroid-resistant/ relapse ITP in China. Patients were randomized to Sitagliptin plus danazol and danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin and Danazol (Experimental): Sitagliptin is given at a dose of 100 mg/m2 qd for 12 weeks. Danazol is given at 200mg bid for 12 weeks.
  Interventions: Drug: Sitagliptin; Drug: Danazol
- Danazol (Active Comparator): Danazol is given at 200mg bid for 12 weeks.
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Sitagliptin — Oral Sitagliptin (100mg/m2 daily) for 12 weeks. DPP4 inhibitors have anti-inflammatory, immunomodulatory, and hematopoietic effects in addition to their glycemic regulatory effects. In vivo experiments found that endogenous DPP-4 inhibits megakaryopoiesis, and knockout or inhibition of DPP4 in vivo can enhance the recovery of hematopoietic function after stress. The loss of DPP-4 activity in DPP-4-/-mice mice resulted in an expansion of the megakaryocyte progenitor population in vivo, the recovery time of platelets was shorter than in normal mice after platelet depletion with anti-mouse CD41 antibody. Compared with ordinary mice, the number of platelets increased, which provides a theoretical basis for the use of DPP-4 inhibitors in patients with ITP, and has potential clinical significance.
  Other Names: JANUVIA
  Arms: Sitagliptin and Danazol
Drug: Danazol — Oral danazol (200 mg twice daily) for 12 weeks.
  Other Names: Danocrine

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of combination of Sitagliptin and danazol versus danazol for the treatment of adults with steroid-resistant/relapse immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 120 adults with steroid-resistant/relapse ITP in China. Patients were randomized to Sitagliptin plus danazol and danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia; Platelet count of less than 30×109/L at enrollment; Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation; 18 years older;

Exclusion Criteria:

Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus) Congestive heart failure Severe arrhythmia Nursing or pregnant women Aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria Creatinine or serum bilirubin levels each 1•5 times or more than the normal range Active or previous malignancy Unable to do blood routine test for the sake of time, distance, economic issues or other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up. Interim analysis was scheduled at 50% through recruitment.

SECONDARY OUTCOMES:
Complete remission | 6 months
  The number of participants (responders) with platelet count>=100x10^9/L (CR) and the absence of bleeding.
Partial remission | 6 months
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) without the administration of any other platelet increasing therapy.
Time to response | 6 months
  Time to response was defined as the time from starting treatment to the time to achieve the response.
Duration of response | 6 months
  Duration of response was measured from the achievement of response to the loss of response.
Incidence of treatment-emergent adverse events | 6 months
  Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-hui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China